CLINICAL TRIAL: NCT04968405
Title: Analysis of the Performance and Safety of the Catalyst CSR Shoulder System - A Prospective Study
Brief Title: Catalyst CSR Shoulder System for Semi or Total Shoulder Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catalyst OrthoScience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1226-9272-01
Record Dates: First submitted 2020-03-11; First posted 2021-07-20 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Osteoarthritis Shoulder; Avascular Necrosis of the Head of Humerus; Rheumatoid Arthritis Shoulder
Keywords: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis; Post-traumatic Arthritis; Correction of functional deformity
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Catalyst CSR Shoulder System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Arm (Other): Intervention with a 510k cleared shoulder arthroplasty device
  Interventions: Device: Catalyst CSR Total Shoulder System

INTERVENTIONS:
Device: Catalyst CSR Total Shoulder System — The Catalyst CSR Shoulder System is a bone preserving total shoulder prosthesis designed for use in patients where the humeral head, neck and glenoid vault are of sufficient bone stock and there is an intact or reconstructable rotator cuff. The design requires minimal bone resection, thus giving the patient an alternative to other total shoulder designs where more bone is removed.

SUMMARY:
Evaluation of the performance and safety of the Catalyst CSR Shoulder System with clinical and radiographic results at multiple time points through 24 months postoperatively This study will be a prospective multi-center study conducted in the United States.

DETAILED DESCRIPTION:
The purpose of this study is to assess the performance and safety of the Catalyst CSR Shoulder System in skeletally mature patients with degenerative disease of the glenohumeral joint where hemi or total shoulder arthroplasty is determined by the surgeon to be the preferred method of treatment. Patients who sign informed consent and meet the inclusion/exclusion criteria will have the Catalyst CSR Shoulder system implanted at participating sites. Data will be collected at baseline (pre-operative), perioperatively, and postoperatively at 3 months, 6 months, 12 months and 24 months. This study is expected to take 36 months to complete.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patient must be skeletally mature with degenerative disease of the glenohumeral joint where hemi or total shoulder arthroplasty
* Meets the Catalyst CSR Shoulder System Indications for Use according to approved labeling

Exclusion Criteria

* Has a history of open surgery to index shoulder prior to treatment with the Catalyst CSR system? (history of previous arthroscopic surgery allowed)
* Has a full thickness rotator cuff tear diagnosed by MFI or marked posterior glenoid wear
* Patient is unwilling or unable to comply with the post-operative care instructions, attend follow visits per the study schedule and complete the study assessments (i.e., Pros)
* The patient is a non-English speaker
* In the opinion of the investigator, is it not in the patient's best interest to participate in this study
* Local or systemic infection, or osteomyelitis of the proximal humerus or scapula; if a systemic infection or a secondary remote infection is suspected or confirmed, joint replacement surgery should be delayed until infection is resolved
* Inadequate or malformed bone that precludes adequate support of fixation of the prosthesis
* Osteoporosis
* Neuromuscular disorders that do not allow control of the joint
* Chronic instability, chronic dislocation or deficient soft tissues and other support structures (e.g., brachial plexus or deltoid muscles)
* Vascular insufficiency
* Subject's age, weight or activity level cause the surgeon to expect early failure of the system
* The patient is unwilling to comply or unable to comply with the post-operative care instructions
* Alcohol, drug, substance abuse or other conditions that would affect or impair the patient from complying with post-operative instructions
* Patients with known sensitivity to Co-Cr-Mo alloys typically used prosthetic devices
* Any disease that could adversely affect the function or expected longevity of the implants (e.g., metabolic disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Assessment Questionnaire | 12 Months
  Change from baseline in patient reported outcome scores using the ASES

SECONDARY OUTCOMES:
Radiographic Assessment | 3 months, 6 months, 12 months, 24 months
  Lack of radiographic evidence of osteolysis, stress shielding or lucent line formation through a minimum of 12-months post operation.
Range of Motion Assessment | Baseline, 3 months, 6 months, 12 months, 24 months
  Change active range of motion (ROM) from baseline (preoperative)
American Shoulder and Elbow Surgeons (ASES) Assessment Questionnaire | Baseline 3 months, 6 months, 12 months, 24 months
  Change from baseline in patient reported outcome scores using the ASES
PROMIS Physical and Mental Function (PROMIS GLOBAL-10) Questionnaire | Baseline 3 months, 6 months, 12 months, 24 months
  Change from baseline in patient reported outcome scores using the PROMIS
Single Assessment Numeric Evaluation (SANE) | Baseline 3 months, 6 months, 12 months, 24 months
  Change from baseline in patient reported outcome scores using the SANE
Visual Analog Score (VAS) Scale | Baseline 3 months, 6 months, 12 months, 24 months
  Change from baseline in patient reported outcome scores using the VAS
Patient Satisfaction Assessment | 6, 12 and 24 months
  Patient Satisfaction

OTHER OUTCOMES:
Patient Safety | perioperatively, 3, 6, 12 and 24 months
  Report of adverse events/serious adverse event rates related to the procedure or device
  * Implant removal rate
  * Revision rate

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Wiater, MD, Principal Investigator — Beaumont Hospital Royal Oak
Locations (3):
- United States (3):
  - Beaumont Hospital Royal Oak, Royal Oak, Michigan
  - Kaiser Permanente Northwest Center for Health Research, Portland, Oregon
  - Lifespan/University Orthopedics, Providence, Rhode Island